CLINICAL TRIAL: NCT04836676
Title: Clinical Validation of C-REX Device for Adaptive Anastomoses: A Multicentre Non-Randomised Controlled Study for Post-Market Clinical Follow-up
Brief Title: Clinical Validation of C-REX Device for Adaptive Anastomoses
Acronym: C-REX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Carponovum AB (Industry)
Collaborators: Stockholm South General Hospital (Other); Karolinska University Hospital (Other); Danderyd Hospital (Other); Capio Sankt Görans Hospital (Other); Ersta Diakoni (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CREX-006
Record Dates: First submitted 2021-03-19; First posted 2021-04-08 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Cancer Colonic
Keywords: Adaptive anastomoses; C-REX; Colorectal cancer; Post-Market
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- C-REX group (Experimental): After resection of the disease in colon, the intestinal ends will be anastomosed by the investigational device, i.e. C-REX LapAid Cath or C-REX RectoAid Cath.
  Interventions: Device: C-REX Device

INTERVENTIONS:
Device: C-REX Device — The investigational devices are C-REX LapAid Cath or C-REX RectoAid Cath. C-REX LapAid Cath consists of an invasive surgical part, i.e. anastomotic ring comprised of two LapAn coupled by DMC/DM, intended for short-term use, and surgical instruments for assisting the placement of the anastomotic ring to intestine.
  C-REX RectoAid Cath consists of an invasive surgical part, i.e. an anastomotic ring comprised of RectoAn and LapAn, intended for short-term use, and surgical instruments for assisting the placement of the anastomotic ring to intestine.
  C-REX LapAid Cath and C-REX RectoAid Cath are easy to use, with unique possibility to control and validate the integrity of the anastomosis during and after surgery.

SUMMARY:
In colorectal surgery, hand suturing and stapling are routine methods for performing intestinal anastomoses, and these methods appear to be similar in terms of clinical safety. Despite several years of experience with surgical procedures as well as improvements to the medical devices, problems with disturbed anastomotic healing leading to leakage and stenosis after colorectal surgery remain a significant challenge for surgeons. A frequency of anastomotic leakage after stapling or suturing has been reported to range from 3% to 20%. In addition, preoperative radiotherapy has been shown to increase the risk of anastomotic leakage even further.

The methods that are used today to detect leakages are unfortunately inaccurately and limited to monitoring symptoms, temperature, CRP-levels, and performing abdominal examinations and CT-scans. These clinical signs and parameters usually become apparent several days after onset of the leakage, which leads to a delayed diagnosis. Anastomotic leakage is not only a significant cause of increased morbidity of complications and mortality in patients, but also associated with increased risk of local recurrence and poor prognosis. Moreover, when reoperation is required to fix the leakage, a permanent stoma may be made at the level of the sigmoid colon and this procedure impacts live quality of patients negatively.

Based on the above considerations, a novel, adaptive anastomotic method has been developed by CarpoNovum to achieve a safer anastomosis. The method's working name is C-REX Ring-locking Procedure. C-REX is referred to our Colorectal anastomotic rings for Re-join the intestinal ends and validate the anastomosis, with function of Extract samples for analysis and conduct X-ray through connected catheters.

The newly developed adaptive anastomotic medical devices, C-REX LapAid Cath and C-REX RectoAid Cath are easy to use, with unique possibility to control the anastomosis during and after surgery. The previous successful pre-market data support a successful CE marking of the devices, which encourages a post-market clinical follow-up (post CE mark clinical study) in patients undergoing colonic resection to collect post-market data of C-REX LapAid Cath and C-REX RectoAid Cath for the purpose of clinical evaluation and risk analysis.

DETAILED DESCRIPTION:
OVERALL DESIGN:

The study is a post-market multicentre non-randomized controlled study. In each investigational site, the investigational personnel shall start with colonic resections, first 10 patients. When surgeons feel confident using the device and ward personal feel confident treating the patient postoperatively, they will initiate rectal resections.

Eligible patients for C-REX LapAid Cath are those requiring resection of the left colon (descending colon and sigmoid) or above the upper rectum (> 15 cm above the anal rim) due to malign or benign disease. Eligible patients for C-REX RectoAid Cath are those requiring resection of the rectum due to malign or benign disease. The proximal limit is upper rectum (< 15 cm above the anal rim) and the distal limit is the anal sphincter.

Patients will be enrolled in the study after they have provided informed consent, having undergone physical examination and been found to meet inclusion criteria. Bowel cleansing prior surgery should be performed according to local routines. The intestinal resection and anastomosis with the investigational devices, i.e. C-REX LapAid Cath or C-REX RectoAid Cath, shall be performed in line with standard procedure of proctocolectomy during hospitalization. Surgeons can utilize catheters that allow monitoring of the anastomosis during and after surgery.

The healing period is expected to be approximately 10 ± 2 days. The short-term implant detaches via necrosis on the inner part of the intestinal surface and is expelled the natural way. The patient can be discharged before expelling of the short-term implant upon investigator's discretion.

The patients will be followed up according to local procedure subsequently. The LARS score shall be assessed at 12 months, and healthcare utilization shall be assessed at 12 months postoperatively.

SUBJECTS:

The aim of this study is to collect post-market data of C-REX LapAid Cath and C-REX RectoAid Cath for the purpose of clinical evaluation and risk analysis. No control group is included in this study.

Considering that similar anastomotic devices have been used in clinic for decades, the study will include about 200 subjects from at least 3 different sites/hospitals. In which, colonic resections shall be applied in 100 subjects, and recta resections in another 100 subjects. The device used is either C-REX LapAid Cath or C-REX RectoAid Cath.

QUALITY CONTROL:

1. Authorization to apply investigational devices:

   According to CarpoNovum's regulation, clinical investigators must be authorized to perform adaptive anastomosis with C-REX LapAid Cath or C-REX RectoAid Cath by performing at least one tutor-led surgery on pigs and at least one train-in surgery on patients with the trainer. When the clinical investigator is authorized to use the investigational devices, he or she receives a certificate.
2. Investigation site selection:

   Investigation sites will be identified to participate in the study based on current experience, referrals from the principle investigator, and training in the use of the investigational devices according to the procedure of surgeon accreditation, and in accordance with ICH GCP guidelines and ISO 14155. It is expected that the surgeons will adhere to and follow protocol of performing adaptive anastomosis provided in the IFUs, and relevant study documents.
3. Monitoring:

   To ensure that the study is appropriately conducted, there is a need for on-site monitoring before, during and after the clinical study. Remote monitoring without visiting the site may be performed as well. The study will be monitored by CarpoNovum or its authorized representatives in accordance the internal procedures of CarpoNovum. The frequency of the visit will be determined by the sponsor and scheduled based on enrolment and the number of active follow-up visits at each site.

   The responsible monitor will evaluate and summarize the results of each monitoring visit in a written report. The reports will be sent to the sponsor and the principal clinical investigators.
4. Traceability and device accountability:

The investigational devices stored in the investigation site in a locked cabin are only accessible to investigation personnel.

The size of the device used in surgery should be recorded in CRF, the Patient Record Label on the device should be pasted on CRF as well. If more than one set of investigational devices are opened during surgery, all Patient Record Labels should be pasted on CRF and reasons for why the devices have been opened during surgery should be recorded.

After surgery, the information of used or opened devices should be noted in Device Accountability. The used investigational devices or opened but not used devices, together with expelled short-term implants should be collected and saved in the investigation site. All components of devices, no matter if they have been used or not, as well as expelled short-term implants if possible, should be hand over to the sponsor when the study is finished. No component of investigational devices should be disposed or lost.

DOCUMENTATION AND DATA MANAGEMENT:

The following information should be clearly documented in medical record of subjects:

* That the subject is informed about the study and that the subject has signed the informed consent forms.
* That the subject is participating in the study; the identification code for the subject, the name of the study, and the study number.
* Which treatment the study refers to.
* Name of clinical investigator.
* All AEs and device deficiencies.

The personal data obtained in the course of the study, in accordance with the informed consent, and in particular clinical findings are subjected to confidentiality. All generated and processed data during the study are protected by subject's identification code. Subjects will also provide his/her written approval for concerned investigation personnel, representatives of the sponsor, monitor and the medical inspection authority, Swedish or foreign, to obtain access to subjects' medical records, to compare them to collected data or reported information. This approval will be granted with reservations that information concerning subjects that become available is not pursued further. Subjects must also give his/her written approval that the study results that concern the subjects can be used in reporting on the study as a whole, provided that no records are pursued further.

For each subject enrolled, regardless of medical device initiation, a CRF must be completed and signed by corresponding study personnel. This applies to those subjects who fail to complete the study. If a subject withdraws from the study, the reason must be noted on CRF.

Data and information of subjects derived from the study, for instance medical records, imagine reports, surgical notes etc. are considered as source data. To ensure that all data are complete and correct, source data verification (SDV) will be confirmed by the monitor.

Comments in CRF should be made with a ballpoint pen with permanent ink in paper based CRF.

In both paper-based CRF and eCRF, if comments are missing in CRF, reasons for this must be stated. No questions, squares, fields or similar should be left without comments.

The responsible clinical investigator is obliged to keep the subject identification lists with the subject's identification code and identity in a safe place at the investigation site, accessible only to the investigation personnel. These source data and subject identification lists will be saved for 10 years after the close of the study at the medical institution.

EARLY STUDY TERMINATION:

CarpoNovum reserves the right to terminate a non-preforming site. Reasons for considering early termination or suspension of an individual site may include, but are not limited to:

* Non-compliance with study protocol or failure to comply with government or local regulations.
* Failure to submit data in a timely manner.
* Failure to comply with or act upon findings.
* Failure to enrol an adequate number of subjects.
* Other reasons mentioned in the PMCIP, including that other investigation sites have enrolled a sufficient number of evaluable subjects which meets the statistical requirements

CarpoNovum reserves the right to discontinue the study at any time due to, but not limited to:

* Strategic considerations of CarpoNovum.
* Force majeure event which results that the study cannot continue.

Upon early termination of the study, the sponsor will notify each investigator immediately at the time of such a decision. Formal documentation will be provided to the Swedish Ethical Review Authority and investigation sites. After such a decision, the investigators must contact all participating subjects to notify them of this decision and its impact on their follow-up.

STATISTICAL CONSIDERATION:

Basic demographic and other baseline characteristics will be analysed for all patients. Summary statistics (arithmetic mean and standard deviation / median and interquartile range, minimum and maximum for quantitative variables, as appropriate) will be presented for the total study population. Frequency tables for qualitative data will be provided. Any deviation from specified statistical plan will be in addition to "per protocol" analysis and will be reported as such.

Any deviations from the specified statistical analysis plan will be described in the study report.

Analysis populations:

ITT (Intention to treat) analysis set - all included researchers who have undergone surgery so that they have been exposed to a risk of leakage according to the primary study point, including those who withdraw or are excluded during the operation or are excluded during follow-up. The primary analysis is based on this analysis set.

Safety analysis set - all researchers who have undergone surgery. Safety endpoints are analyzed with this analysis set.

Per protocol analysis set - all researchers who completed the study without protocol deviations. As a secondary analysis, the primary analysis is also performed on this analysis set.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age ≥ 18 years old.
2. Planned resection due to benign or malign disease in the left colon or the rectum.
3. Cognitive ability to take part in the study and understand the information the patient receives about participating in the study and provide informed consent.

Exclusion Criteria:

1. Pre-existing health conditions requiring surgery, such as intestinal obstruction or perforation, local or systemic infections, peritonitis, or intestinal ischemia.
2. Non-curable metastatic disease (cancer with multi-organ metastases).
3. Intestinal or anal stenosis or other obstructions distal to the anastomotic site.
4. Contraindications to general anaesthesia.
5. Other conditions upon surgeon's discretion that may warrant exclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of radiologically verified clinical anastomotic leakage related to the investigational device(s). | Up to 30 days after surgery
  Anastomotic leakage is defined as a defect in the intestinal wall at the site of the anastomosis (including C-REX short-term implants) which leads to a communication between the intra- and extraluminal spaces. The severity of anastomotic leakage should be classified according to the clinically required measures. Grade A anastomosis leakage does not lead to any change in the researcher's handling, while Grade B leakage requires active therapeutic intervention but is manageable without relaparotomy. Grade C anastomotic leakage requires relaparotomy.

SECONDARY OUTCOMES:
Air leak test during surgery | During surgery
  Negative result of air leak test during surgery
C-REX integrity pressure test (optional) | During surgery
  To confirm that the two anastomotic rings are properly locked to each other, measure integrity pressure through catheters connected to DMC (if DMC is applied). By infusing air into the closed space adjacent to the anastomosis via on catheter and concomitantly camping the other three catheters. When the pressure in the closed space exceeds the contact-induced closure by the joined intestinal segments, the pressure abruptly dropped and is defined as integrity pressure
Duration of surgery | During surgery
  The time to complete the operation
Time to evacuation of the short-term implant | About 10 ± 2 days after surgery
  The subject informs the clinical investigator and hand over the expelled short-term implant
Postoperative complication assessment | Up to 30 days after surgery
  The clinical investigator visits the subject every day after surgery up to evacuation of the short-term implant or the subject has been discharged from the hospital, and examines the subjects and assesses postoperative complications according to Clavien-Dindo classification.
Postoperative bowel dysfunction assessment | At 12 months post-surgery
  Postoperative bowel dysfunction assessment according to low anterior resection syndrome (LARS) assessment at 12 months post-surgery.
Healthcare utilization patterns assessment | At 12 months post-surgery
  To assess healthcare utilization patterns in patients who have undergone surgery with investigational devices
Incidence rate of investigational device(s) related adverse event (AE) and serious adverse event (SAE) other than anastomotic leakage | Up to 12 months after surgery
  Any investigational device(s) related adverse event (AE) and serious adverse event (SAE) other than anastomotic leakage

OTHER OUTCOMES:
Assessment of post-operative satisfaction | Through study process, an average of 3 months
  Assessment of post-operative satisfaction with the investigational device and educational material evaluation in investigational personnel after ±10 C-REX surgeries by a surgeon by a questionnaire comprising both multiple-choice questions on a 5-point Likert scale and open-ended questions for qualitative investigation.

CONTACTS AND LOCATIONS:
Overall Officials: Torbjörn Holm, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (5):
- Sweden (5):
  - Danderyds Sjukhus, Danderyd, Stockholm County
  - Capio Saint Göran's Sjukhus, Stockholm
  - Ersta diakoni, Stockholm
  - Södersjukhuset, Stockholm
  - Karolinska Universitetssjukhuset, Stockholm